CLINICAL TRIAL: NCT07349277
Title: Evaluation of sFlt-1/PlGF Ratio, Osteoprotegerin (OPG) and Soluble Endoglin (sEng) as Predictive Biomarkers in the Diagnosis and Treatment Evaluation of Preeclampsia
Brief Title: Evaluation of sFlt-1/PlGF Ratio ,OPG and sEng as Predictive Biomarkers in the Diagnosis and Treatment Evaluation of Preeclampsia
Acronym: PE-POSS
Status: Recruiting | Type: Observational
Sponsor: Ammar Jassim Abed (Other)
Responsible Party: Sponsor-Investigator, Ammar Jassim Abed, Master's Student (MSc Researcher), Principal Investigator, University of Thi-Qar
Organization: University of Thi-Qar (Other)
Other Study IDs: 35918
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Preeclampsia; Gestational Hypertension; Hypertensive Disorders of Pregnancy
Keywords: sFlt-1/PlGF ratio; Soluble Endoglin (sEng); Osteoprotegerin (OPG); Angiogenesis; Placental Dysfunction; Preeclampsia; methyldopa
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples (5 mL each) will be collected from three groups of pregnant women:
  Women diagnosed with preeclampsia who are not receiving antihypertensive treatment.
  Women diagnosed with preeclampsia who are receiving antihypertensive treatment.
  Healthy pregnant women as control subjects.
  Serum will be separated by centrifugation and aliquoted into two tubes for storage. All samples will be frozen at -80°C for future biomarker analysis.
  Retained biospecimens will include serum samples only. Samples will be labeled with anonymized participant codes to protect privacy. They may be used for measurement of angiogenic and anti-angiogenic biomarkers (sFlt-1, PlGF, soluble endoglin, and osteoprotegerin)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Preeclampsia - No Antihypertensive Treatment: This group includes pregnant women diagnosed with preeclampsia. Blood samples are collected at the time of diagnosis before starting any antihypertensive treatment. All participants will receive standard clinical care after sample collection. Samples will be processed, aliquoted, and stored at -80°C for biomarker analysis (sFlt-1, PlGF, soluble endoglin, and osteoprotegerin).
- Preeclampsia - With Antihypertensive Treatment: is group includes pregnant women diagnosed with preeclampsia who are receiving standard antihypertensive therapy as part of their clinical care. Blood samples (5 mL) will be collected for measurement of biomarkers (sFlt-1, PlGF, sEng, OPG). Samples will be processed, aliquoted, and stored at -80°C. Clinical parameters and treatment details will also be recorded for analysi
- Healthy Pregnant Controls: his group includes healthy pregnant women without preeclampsia. Blood samples (5 mL) will be collected to serve as controls for biomarker analysis. Samples will be processed, aliquoted, and stored at -80°C. Participants will receive routine prenatal care.

SUMMARY:
his study investigates the effectiveness of three specific biological markers (biomarkers) in the blood-the sFlt-1/PlGF ratio, soluble endoglin (sEng), and osteoprotegerin (OPG)-to better diagnose and monitor preeclampsia. Preeclampsia is a serious pregnancy complication characterized by high blood pressure and potential organ damage that affects 2-8% of pregnancies worldwide

DETAILED DESCRIPTION:
Preeclampsia is a pregnancy-specific hypertensive disorder characterized by newonset hypertension and proteinuria or other maternal organ dysfunction after 20 weeks of gestation. It affects 2-8% of pregnancies globally and remains a major contributor to maternal and perinatal morbidity and mortality The etiology is multifactorial, but placental dysfunction and abnormal angiogenesis are central to its pathogenesis. Given the limitations of current clinical indicators (e.g., blood pressure, proteinuria), there is growing interest in identifying predictive and diagnostic biomarkers to improve early detection, prognosis, and monitoring of therapeutic response. This study proposes to investigate three biomarkers: the sFlt-1/PlGF ratio, soluble endoglin (sEng), and osteoprotegerin (OPG), based on their roles in angiogenesis and endothelial dysfunction, which are hallmarks of preeclampsia

sFlt-1/PlGF Ratio Soluble fms-like tyrosine kinase-1 (sFlt-1) is an anti-angiogenic protein that binds to vascular endothelial growth factor (VEGF) and placental growth factor (PlGF), preventing their interaction with endothelial receptors. The imbalance, especially elevated sFlt-1 and decreased PlGF, is characteristic of preeclampsia. Numerous studies, including the multicenter PROGNOSIS trial, have validated the sFlt-1/PlGF ratio as a strong predictor of preeclampsia. A ratio ≥85 is associated with a high risk of developing preeclampsia within two weeks, while ≤38 effectively rules it out .

Soluble Endoglin (sEng) Endoglin is a co-receptor for transforming growth factor-beta (TGF-β), involved in vascular development. Its soluble form (sEng) acts as a decoy receptor, inhibiting TGF-β signaling, contributing to endothelial dysfunction, a key feature of preeclampsia. sEng levels are elevated in the maternal circulation prior to clinical onset and correlate with disease severity.

Osteoprotegerin (OPG) OPG, a member of the TNF receptor superfamily, is primarily involved in bone metabolism but also plays a role in vascular biology. Some studies have reported altered OPG levels in preeclampsia, potentially reflecting vascular damage or endothelial activation . Its role remains less defined, but it may complement other angiogenic markers in profiling disease status.

ELIGIBILITY:
IInclusion Criteria:

* Pregnant women between 20 and 36 weeks of gestation
* Age between 18 and 45 years
* Attending the antenatal clinic at the study site

Exclusion Criteria:

* Chronic hypertension
* Renal disease
* Diabetes mellitus
* Multiple gestations
* Autoimmune disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: he study population will include pregnant women aged 18-45 years, between 20 and 36 weeks of gestation, attending the antenatal clinic at the study site. Participants will be divided into three groups:
  Pregnant women diagnosed with preeclampsia who have not yet received antihypertensive treatment.
  Pregnant women diagnosed with preeclampsia who are receiving antihypertensive treatment.
  Healthy pregnant women serving as control subjects.
  Exclusion criteria include pre-existing chronic hypertension, renal disease, diabetes mellitus, multiple gestations, or autoimmune disorders.
  All participants will provide informed consent before enrollment. Blood samples will be collected for biomarker analysis (sFlt-1, PlGF, soluble endoglin, and osteoprotegerin). This population has been selected to allow comparison of biomarker levels in different clinical scenarios and to evaluate their
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Serum sFlt-1 concentration | At enrollment (20-36 weeks of gestation)
  Measurement of serum sFlt-1 levels in maternal serum using ELISA
Serum PlGF concentration | At enrollment (20-36 weeks of gestation)
  Measurement of serum placental growth factor (PlGF) levels in maternal serum using ELISA.
sFlt-1/PlGF ratio | At enrollment (20-36 weeks of gestation)
  Calculated ratio of serum sFlt-1 to serum PlGF concentrations
Serum Osteoprotegerin (OPG) concentration | At enrollment (20-36 weeks of gestation)
  Measurement of serum osteoprotegerin (OPG) levels in maternal serum using ELISA.
Serum sENG(Souble Endoglin) concentration | At enrollment (20-36 weeks of gestation)
  Measurement of serum soluble endoglin (sENG) levels in maternal serum using ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- Bint Al Huda Maternity Hospital, Nasiriyah, Dhi Qar, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Yes - De-identified individual participant data (IPD) will be available upon reasonable request to qualified researchers. Data will include biomarker measurements (sFlt-1, PlGF, sEng, OPG) and relevant clinical parameters. Requests will be reviewed by the principal investigator, and shared under a data use agreement ensuring confidentiality. Data will be available 12 months after publication of the study results.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified individual participant data (IPD) will be made available to qualified researchers upon reasonable request. Supporting information to be shared includes the study protocol, statistical analysis plan (SAP), and analytic code. Data will be provided in an anonymized format, with requests reviewed by the principal investigator and shared under a data use agreement ensuring confidentiality. Data will be available 12 months after publication of the study results.

REFERENCES:
- [Background] Brown MA, Magee LA, Kenny LC, Karumanchi SA, McCarthy FP, Saito S, Hall DR, Warren CE, Adoyi G, Ishaku S; International Society for the Study of Hypertension in Pregnancy (ISSHP). The hypertensive disorders of pregnancy: ISSHP classification, diagnosis & management recommendations for international practice. Pregnancy Hypertens. 2018 Jul;13:291-310. doi: 10.1016/j.preghy.2018.05.004. Epub 2018 May 24. No abstract available. PMID 29803330
- [Background] Miller JJ, Higgins V, Melamed N, Hladunewich M, Ma L, Yip PM, Fu L. Clinical Validation of the sFlt-1:PlGF Ratio as a Biomarker for Preeclampsia Diagnosis in a High-Risk Obstetrics Unit. J Appl Lab Med. 2023 May 4;8(3):457-468. doi: 10.1093/jalm/jfad003. PMID 36869760
- [Background] Zeisler H, Llurba E, Chantraine F, Vatish M, Staff AC, Sennstrom M, Olovsson M, Brennecke SP, Stepan H, Allegranza D, Dilba P, Schoedl M, Hund M, Verlohren S. Predictive Value of the sFlt-1:PlGF Ratio in Women with Suspected Preeclampsia. N Engl J Med. 2016 Jan 7;374(1):13-22. doi: 10.1056/NEJMoa1414838. PMID 26735990
- [Background] Venkatesha S, Toporsian M, Lam C, Hanai J, Mammoto T, Kim YM, Bdolah Y, Lim KH, Yuan HT, Libermann TA, Stillman IE, Roberts D, D'Amore PA, Epstein FH, Sellke FW, Romero R, Sukhatme VP, Letarte M, Karumanchi SA. Soluble endoglin contributes to the pathogenesis of preeclampsia. Nat Med. 2006 Jun;12(6):642-9. doi: 10.1038/nm1429. Epub 2006 Jun 4. PMID 16751767